CLINICAL TRIAL: NCT06499571
Title: G.A.L.T.O.S. Geographic Atrophy Long-Terms Outcomes Study: An Ambispective Noninterventional Study to Describe the Patient Demographics and Outcomes of Patients With Geographic Atrophy (GA) Secondary to AMD in Clinical Practice
Brief Title: Geographic Atrophy Long-Terms Outcomes Study
Acronym: GALTOS
Status: Completed | Type: Observational
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: GAL-21-NIS
Record Dates: First submitted 2024-04-23; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Geographic Atrophy
Keywords: GA Outcomes
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Geographic Atrophy (GA ) : GA (both eyes with GA)
- Cohort 2: GA : nAMD (1 eye with GA; the other eye with nAMD, including MNV)
- Cohort 3: GA : early/intermediate AMD (1 eye with GA; the other eye with early/intermediate AMD)
  o Other subgroups (GA : drusen, GA : reticular pseudodrusen) will be consider if the sample size allows AMD: Age -Related Macular Degeneration MNV: Macular Neovascularization nAMD: Neovascular Age -Related Macular Degeneration

SUMMARY:
The purpose of this study is to describe functional and long-term clinical outcomes of patients with a diagnosis of Geographic Athrophy secondary to Age related Macular Degenaration in Clinical Practice

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients:

* Aged 60 years or over at the time of GA diagnosis
* Patients providing informed consent to participate in the study; if the patient is physically incapable of completing the electronic consent form, the form can be completed by a legally acceptable representative of the patient (including an impartial witness, where required)
* Patients first diagnosed with GA in at least 1 eye between 3 and 10 years prior to index date
* For patients with unilateral GA, the other eye should show signs of AMD (i.e., the non-GA eye should present with at least drusen, reticular pseudodrusen, or wet-AMD)

Inclusion criteria for caregivers:

* Aged 18 years or over at the time of consent
* Caregivers who self-identify as the primary caregiver for a patient for whom documented informed consent for inclusion in the study has been obtained

Exclusion Criteria:

Exclusion criteria for patients:

* Patients diagnosed with GA due to causes other than AMD (e.g., monogenetic macular dystrophies [Stargardt disease, other], toxic maculopathies) in either eye
* GA with any concurrent intraocular condition that in the opinion of the treating physician would require surgical or intravitreal intervention (for the prevention or treatment of visual loss) during the study or might impact the interpretation of routine clinical assessments e.g., glaucoma, cataract, proliferative diabetic retinopathy. Patients first diagnosed with GA less than 3 years prior to the date of consent
* Patients who have not attended a healthcare institution for the management of GA following diagnosis of GA (a minimum of 2 routine clinical visits for monitoring of GA that included assessment of at least BCVA should be documented in the medical records)
* Patients who have been enrolled in an interventional clinical trial in which they received medication for any retinal condition (note: patients with bilateral GA should be excluded only if both eyes received the pharmacological intervention)

Exclusion criteria for caregivers:

* Caregivers for whom documented informed consent has not been obtained for participation in the GALTOS survey
* Caregivers with any significant mental incapacity that would prevent them from participating in the survey
* Paid caregivers

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received a diagnosis of GA between 3 and 10 years prior to enrollment across 22 ophthalmology centers in Australia, Canada, France, Germany, Italy, and UK.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in GA total area size | Through study completion; between 4 and 11 years
  Mean GA total area size and Mean change in GA total area size
Change from baseline in BCVA | Through study completion; between 4 and 11 years
  Mean BCVA and Mean change in BCVA
Percentage of participants with visual impairment/blindness | Through study completion; between 4 and 11 years
  Percentage of participants with moderate/severe visual impairment or blindness
Percentage of participants with microperimetry assessment | Through study completion; between 4 and 11 years
  Percentage of participants with any microperimetry assessments since GA diagnosis
Mean change in functional parameters in patients with microperimetry assessments | Through study completion; between 4 and 11 years
  Mean/Median and Mean change in retinal sensitivity.
Mean change in functional parameters in patients with microperimetry assessments | Through study completion; between 4 and 11 years
  Mean/Median and Mean change in fixation stability.
Mean change in functional parameters in patients with microperimetry assessments | Through study completion; between 4 and 11 years
  Mean/Median and Mean change in number of scotoma points.
Percentage of eyes with disease progression | Through study completion; between 4 and 11 years
  Percentage of eyes that complete any of the protocol-defined disease progression trajectories and Mean time from GA diagnosis to disease progression

SECONDARY OUTCOMES:
Proportion of GA eyes with presence of selected characteristics | Through study completion; between 4 and 11 years
  Proportion of GA eyes with presence of any of the following: nAMD, drusen, pseudodrusen, foveal involvement, unifocal/multifocal GA, hypopigmentation
Proportion of non-GA eyes with presence of AMD | Through study completion; between 4 and 11 years
  Proportion of non-GA eyes with presence of any of the following: early/intermediate AMD, nAMD, MNV
Mortality rate | From enrollment until end of follow-up; 12 (+6) months after the follow-up period.
  Mortality rate during study follow-up
GA-related HCRU during the observation period | Through study completion; between 4 and 11 years
  Number of medical visits (outpatient, low vision clinic, etc.)
GA-related HCRU during the observation period | Through study completion; between 4 and 11 years
  number of imaging tests (F, A, FAF, CFP, OCT, OCTA, etc.)
GA-related HCRU during the observation period | Through study completion; between 4 and 11 years
  number of prescribed vision aids, per participant
Patient-reported HRQoL | From enrollment until end of follow-up; 12 (+6) months after the follow-up period.
  Score of the EQ-5D.
Patient-reported HRQoL | From enrollment until end of follow-up; 12 (+6) months after the follow-up period.
  Score of the HADS
Patient-reported HRQoL | From enrollment until end of follow-up; 12 (+6) months after the follow-up period.
  Score of the AQoL-7D for Australian sites only.
Patient-reported performance | From enrollment until end of follow-up; 12 (+6) months after the follow-up period.
  Scores/answers to the NEI-VFQ-25 questionnaire.
Patient-reported performance | From enrollment until end of follow-up; 12 (+6) months after the follow-up period.
  Scores/answers to the GALTOS survey.
Assisted-care patient journey | From enrollment until end of follow-up; 12 (+6) months after the follow-up period.
  Proportion of patients requiring support from an informal caregiver, receiving assisted care at home or in assisted living
Assisted-care patient journey | From enrollment until end of follow-up; 12 (+6) months after the follow-up period.
  mean/median time from GA diagnosis to first type of assistance
Financial impact of GA on patients and caregivers | From enrollment until end of follow-up; 12 (+6) months after the follow-up period.
  Selected items of the GALTOS survey (including the cost, in the past 12 months, associated to prescriptions, assistive devices, healthcare-related travel, etc.)
Associations between patient characteristics and disease progression/functional outcomes and/or clinical/anatomical/functional outcome measures | Through study completion; between 4 and 11 years
  Measures of association such as correlation coefficients, chi-square statistic, and potentially coefficients from multivariate analysis methods characterizing the relationships of interest

CONTACTS AND LOCATIONS:
Locations (5):
- Sydney West Retina, Westmead, New South Wales, Australia
- Centre Hospitalier de la Croix Rousse, Lyon, Rhone, France
- Universitaetsklinikum Muenster, Münster, North Rhine-Westphalia, Germany
- Azienda Socio Sanitaria Territoriale Fatebenefratelli (Presidio Ospedale Sacco), Milan, Italy
- Belfast Health & SC Trust, Belfast, United Kingdom

REFERENCES:
- [Background] Fleckenstein M, Mitchell P, Freund KB, Sadda S, Holz FG, Brittain C, Henry EC, Ferrara D. The Progression of Geographic Atrophy Secondary to Age-Related Macular Degeneration. Ophthalmology. 2018 Mar;125(3):369-390. doi: 10.1016/j.ophtha.2017.08.038. Epub 2017 Oct 27. PMID 29110945
- [Background] Sacconi R, Corbelli E, Querques L, Bandello F, Querques G. A Review of Current and Future Management of Geographic Atrophy. Ophthalmol Ther. 2017 Jun;6(1):69-77. doi: 10.1007/s40123-017-0086-6. Epub 2017 Apr 8. PMID 28391446
- [Background] Kandasamy R, Wickremasinghe S, Guymer R. New Treatment Modalities for Geographic Atrophy. Asia Pac J Ophthalmol (Phila). 2017 Nov-Dec;6(6):508-513. doi: 10.22608/APO.2017262. Epub 2017 Sep 14. PMID 28905539
- [Background] Nielsen, MK. Geographic Atrophy. Eyewiki. 2021. Available from: https://eyewiki.org/Geographic_Atrophy.
- [Background] Sastre-Ibanez M, Barreiro-Gonzalez A, Gallego-Pinazo R, Dolz-Marco R, Garcia-Armendariz B. Geographic atrophy: Etiopathogenesis and current therapies. Arch Soc Esp Oftalmol (Engl Ed). 2018 Jan;93(1):22-34. doi: 10.1016/j.oftal.2017.07.004. Epub 2017 Sep 5. English, Spanish. PMID 28886928
- [Background] Boyer DS, Schmidt-Erfurth U, van Lookeren Campagne M, Henry EC, Brittain C. THE PATHOPHYSIOLOGY OF GEOGRAPHIC ATROPHY SECONDARY TO AGE-RELATED MACULAR DEGENERATION AND THE COMPLEMENT PATHWAY AS A THERAPEUTIC TARGET. Retina. 2017 May;37(5):819-835. doi: 10.1097/IAE.0000000000001392. PMID 27902638
- [Background] Kim A, Devine B, Campbell J, Shirneshan E, Zhao C, Bansal A. Healthcare Resource Utilization and Costs in Patients with Geographic Atrophy Secondary to Age-Related Macular Degeneration. Clin Ophthalmol. 2021 Jun 23;15:2643-2651. doi: 10.2147/OPTH.S307603. eCollection 2021. PMID 34188442
- [Background] Daien V, Nguyen V, Essex RW, Guymer R, Arnold JJ, Munk M, Ceklic L, Gillies MC, Barthelmes D; Fight Retinal Blindness! investigators. Prevalence and characteristics of macular atrophy in eyes with neovascular age-related macular degeneration. A study from a long-term observational dataset: the Fight Retinal Blindness! project. Br J Ophthalmol. 2020 Aug;104(8):1064-1069. doi: 10.1136/bjophthalmol-2019-315055. Epub 2019 Dec 16. PMID 31843790
- [Background] Sakurada Y, Yoneyama S, Sugiyama A, Tanabe N, Kikushima W, Mabuchi F, Kume A, Kubota T, Iijima H. Prevalence and Genetic Characteristics of Geographic Atrophy among Elderly Japanese with Age-Related Macular Degeneration. PLoS One. 2016 Feb 26;11(2):e0149978. doi: 10.1371/journal.pone.0149978. eCollection 2016. PMID 26918864
- [Background] Patnaik J, Pecen P, Lynch A, Siringo F, Mathias M, Mandava N. The National Eye Institute Visual Function Questionnaire-25 in Patients with Age-Related Macular Degeneration and Controls. Invest Ophthalmol Vis Sci. 2019;60(9):67-.
- [Background] Sivaprasad S, Tschosik E, Kapre A, Varma R, Bressler NM, Kimel M, Dolan C, Silverman D. Reliability and Construct Validity of the NEI VFQ-25 in a Subset of Patients With Geographic Atrophy From the Phase 2 Mahalo Study. Am J Ophthalmol. 2018 Jun;190:1-8. doi: 10.1016/j.ajo.2018.03.006. Epub 2018 Mar 10. PMID 29530781
- [Background] Patel PJ, Ziemssen F, Ng E, Muthutantri A, Silverman D, Tschosik EA, Cantrell RA. Burden of Illness in Geographic Atrophy: A Study of Vision-Related Quality of Life and Health Care Resource Use. Clin Ophthalmol. 2020 Jan 8;14:15-28. doi: 10.2147/OPTH.S226425. eCollection 2020. PMID 32021065
- [Background] Sivaprasad S, Tschosik EA, Guymer RH, Kapre A, Suner IJ, Joussen AM, Lanzetta P, Ferrara D. Living with Geographic Atrophy: An Ethnographic Study. Ophthalmol Ther. 2019 Mar;8(1):115-124. doi: 10.1007/s40123-019-0160-3. Epub 2019 Jan 31. PMID 30706242
- [Background] Higgins BE, Taylor DJ, Bi W, Binns AM, Crabb DP. Novel computer-based assessments of everyday visual function in people with age-related macular degeneration. PLoS One. 2020 Dec 7;15(12):e0243578. doi: 10.1371/journal.pone.0243578. eCollection 2020. PMID 33284855
- [Background] Singh RP, Patel SS, Nielsen JS, Schmier JK, Rajput Y. Patient-, caregiver-, and eye care professional-reported burden of geographic atrophy secondary to age-related macular degeneration. Am J Ophthalmic Clin Trials. 2019;2(1):1-6. Available from: https://doi.org/10.25259/AJOCT-9-2018
- [Background] Richard AJ, Duker JS, Reichel E. Geographic atrophy: where we are now and where we are going. Curr Opin Ophthalmol. 2021 May 1;32(3):247-252. doi: 10.1097/ICU.0000000000000763. PMID 33741759
- [Background] Halawa OA, Lin JB, Miller JW, Vavvas DG. A Review of Completed and Ongoing Complement Inhibitor Trials for Geographic Atrophy Secondary to Age-Related Macular Degeneration. J Clin Med. 2021 Jun 11;10(12):2580. doi: 10.3390/jcm10122580. PMID 34208067
- [Background] Sunness JS, Margalit E, Srikumaran D, Applegate CA, Tian Y, Perry D, Hawkins BS, Bressler NM. The long-term natural history of geographic atrophy from age-related macular degeneration: enlargement of atrophy and implications for interventional clinical trials. Ophthalmology. 2007 Feb;114(2):271-7. doi: 10.1016/j.ophtha.2006.09.016. PMID 17270676
- [Background] Chakravarthy U, Bailey CC, Johnston RL, McKibbin M, Khan RS, Mahmood S, Downey L, Dhingra N, Brand C, Brittain CJ, Willis JR, Rabhi S, Muthutantri A, Cantrell RA. Characterizing Disease Burden and Progression of Geographic Atrophy Secondary to Age-Related Macular Degeneration. Ophthalmology. 2018 Jun;125(6):842-849. doi: 10.1016/j.ophtha.2017.11.036. Epub 2018 Feb 1. PMID 29366564